CLINICAL TRIAL: NCT01955460
Title: A Pilot Study of Lymphodepletion Plus Adoptive Cell Transfer With TGF-Beta Resistant (DNRII) and NGFR Transduced T-Cells Followed by High Dose Interleukin-2 in Patients With Metastatic Melanoma
Brief Title: Genetically Modified T-Cells Followed by Aldesleukin in Treating Patients With Stage III-IV Melanoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 2012-0758; NCI-2014-01211 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RP110553-P4; RM1012-012-1; 2012-0758 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Melanoma; Stage III Cutaneous Melanoma AJCC v7; Stage IIIA Cutaneous Melanoma AJCC v7; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Cyclophosphamide; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy, autologous T-cell immunotherapy) (Experimental): Patients receive cyclophosphamide IV over 2 hours on days -7 and -6, fludarabine phosphate IV daily over 15-30 minutes on days -5 to -1, and TGFb DNRII-transduced autologous TIL and NGFR-transduced autologous T lymphocytes IV over up to 4 hours on day 0. Patients then receive high-dose aldesleukin IV over 15 minutes every 8-16 hours on days 1-5 (up to 15 doses) and 22-26 (up to 15 doses).
  Interventions: Biological: Aldesleukin; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Biological: NGFR-transduced Autologous T Lymphocytes; Biological: TGFbDNRII-transduced Autologous Tumor Infiltrating Lymphocytes

INTERVENTIONS:
Biological: Aldesleukin — Given IV
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: NGFR-transduced Autologous T Lymphocytes — Given IV
Biological: TGFbDNRII-transduced Autologous Tumor Infiltrating Lymphocytes — Given IV
  Other Names: TGFbDNRII-transduced Autologous TILs

SUMMARY:
This pilot phase I trial studies the side effects and best dose of genetically modified T-cells followed by aldesleukin in treating patients with stage III-IV melanoma. T-cells are a type of white blood cell that help the body fight infections. Genes that may help the T-cells recognize melanoma cells are placed into the T-cells in the laboratory. Adding these genes to the T cells may help them kill more tumor cells when they are put back in the body. Aldesleukin may enhance this effect by stimulating white blood cells to kill more melanoma cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Primary for Cohort A:

I. To assess the feasibility and safety of autologous transforming growth factor beta (TGFb) resistant (DNRII transduced) and NGFR transduced tumor infiltrating lymphocytes (TIL) in patients with metastatic melanoma.

Primary for Cohort B:

I. To assess the feasibility and safety of autologous TGBβ resistant (DNRII transduced) TIL in patients with metastatic melanoma. Feasibility will be defined as the production of virally transduced T cells and treatment of patients with these cells

SECONDARY OBJECTIVES:

Secondary for Cohort A:

I. To determine the survival and immune function of TGFb resistant (DNRII transduced) TIL in vivo.

II. To assess the anti-tumor effects of TGFb resistant (DNRII transduced) TIL.

Secondary for Cohort B:

I. To determine the survival and immune function of TGFβ resistant (DNRII transduced) TIL in vivo

II. To assess the anti-tumor effects of TGFβ resistant (DNRII transduced) TIL.

OUTLINE:

Patients receive cyclophosphamide intravenously (IV) over 2 hours on days -7 and -6, fludarabine phosphate IV daily over 15-30 minutes on days -5 to -1, and TGFb DNRII-transduced autologous TIL and NGFR-transduced autologous T lymphocytes IV over up to 4 hours on day 0. Patients then receive high-dose aldesleukin IV over 15 minutes every 8-16 hours on days 1-5 (up to 15 doses) and 22-26 (up to 15 doses).

After completion of study treatment, patients are followed up at 6 and 12 weeks, every 3 months for 1 year and then yearly for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have metastatic melanoma or stage III in-transit, subcutaneous, or regional nodal disease (Turnstile I)
* Patients must have a lesion amenable to resection or the collection of up to 5 needle core samples for the generation of TIL. (Turnstile I)
* Patients must receive a magnetic resonance imaging (MRI)/computed tomography (CT)/positron emission tomography (PET) of the brain within 6 months of signing informed consent; if new lesions are present, patient must have definitive treatment; principal investigator (PI) or his designee should make final determination regarding enrollment (Turnstile I)
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0-2 within 30 days of signing informed consent (Turnstile I)
* Patients previously treated with immunotherapy, targeted therapy, or no therapy (treatment naive) will be eligible (Turnstile I)
* Patients receiving cytotoxic agents will be evaluated by the PI or his designee for eligibility suitability (Turnstile I)
* Patients with a negative pregnancy test (urine or serum) must be documented within 14 days of screening for women of childbearing potential (WOCBP); a WOCBP has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 12 consecutive months (i.e. who has not had menses at any time in the preceding 12 consecutive months) (Turnstile I)
* Patients must have adequate TIL available (Turnstile II); pre-rapid expansion procedure (Pre-REP) TIL generated in the similar clinical trial 2004-0069 may also be utilized for Turnstile II
* Patients must have at least one biopsiable measurable metastatic melanoma, lesion > or = to 1 cm (Turnstile II)
* Patients may have brain lesions =< 1 cm each; the PI or designee will approve the treatment (Turnstile II)
* Patients of both genders must practice birth control for four months after receiving the preparative regimen (lymphodepletion) and continue to practice birth control throughout the study; patients must have a documented negative pregnancy test (urine or serum) for women who have menstruation in the past 12 months and without sterilization surgery (Turnstile II)
* Unless surgically sterile by bilateral tubal ligation or vasectomy of partner(s), the patient agrees to continue to use a barrier method of contraception throughout the study such as: condom, diaphragm, hormonal, intrauterine device (IUD), or sponge plus spermicide; abstinence is an acceptable form of birth control (Turnstile II)
* Patients with negative pregnancy test (urine or serum) must be documented within 14 days of screening for WOCBP; a WOCBP has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 12 consecutive months (i.e. who has not menses at any time in the preceding 12 consecutive months) (Turnstile II)
* Clinical performance status of ECOG 0-2 within 30 days of signing informed consent (Turnstile II)
* Absolute neutrophil count greater than or equal to 1000/mm^3 (Turnstile II)
* Platelet count greater than or equal to 100,000/mm^3 (Turnstile II)
* Hemoglobin greater than or equal to 8.0 g/dl (Turnstile II)
* Serum alanine aminotransferase (ALT) less than three times the upper limit of normal (Turnstile II)
* Serum creatinine less than or equal to 1.6 mg/dl (Turnstile II)
* Total bilirubin less than or equal to 2.0 mg/dl, except in patients with Gilbert's syndrome who must have a total bilirubin less than 3.0 mg/dl (Turnstile II)
* A stress cardiac test (stress thallium, stress multi gated acquisition scan [MUGA], dobutamine echocardiogram or other stress test that will rule out cardiac ischemia) within 6 months of lymphodepletion (Turnstile II)
* Pulmonary function tests (forced expiratory volume in one second [FEV1] > 65% or forced vital capacity [FVC] > 65% of predicted) within 6 months of lymphodepletion (Turnstile II)
* MRI/CT/PET of the brain within 30 days of lymphodepletion (Turnstile II)

Exclusion Criteria:

* Active systemic infections requiring intravenous antibiotics, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system; PI or his designee shall make the final determination regarding appropriateness of enrollment (Turnstile I)
* Primary immunodeficiency and need for chronic steroid therapy, however prednisone is allowed at < 10 mg/day (Turnstile I)
* Patients who are pregnant or nursing (Turnstile I)
* Presence of a significant psychiatric disease, which in the opinion of the principal investigator or his designee, would prevent adequate informed consent (Turnstile I)
* Has had prior systemic cancer therapy within the past four weeks or v-raf murine sarcoma viral oncogene homolog B (B-RAF) or mitogen-activated protein kinase (MEK) inhibitors within 7 days at the time of the start of the lymphodepletion regimen (Turnstile II)
* Women who are pregnant will be excluded because of the potentially dangerous effects of the preparative chemotherapy on the fetus (Turnstile II)
* Any active systemic infections requiring intravenous antibiotics, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, such as abnormal stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease; PI or his designee shall make the final determination regarding appropriateness of enrollment (Turnstile II)
* Any form of primary or secondary immunodeficiency; must have recovered immune competence after chemotherapy or radiation therapy as evidenced by lymphocyte counts (> 500/mm^3), white blood cell (WBC) (> 3,000/mm^3) or absence of opportunistic infections (Turnstile II)
* Require steroid therapy or steroid-containing compounds, or have used systemic steroids in the past 4 weeks, or have used topical or inhalational steroids in the past 2 weeks prior to lymphodepletion; the exception being patients on chronic physiologic dose of steroid (Turnstile II)
* Presence of a significant psychiatric disease, which in the opinion of the principal investigator or his designee, would prevent adequate informed consent or render immunotherapy unsafe or contraindicated (Turnstile II)
* Patients who are solid organ transplant recipients
* Patients with prior bone marrow or stem cell transplantation

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2014-10-15 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
(Cohort A) Generation of TGF alpha (TGFa)-DNRII and NGFR transduced tumor infiltrating lymphocytes (TILs) | Up to 5 years
  Feasibility of generating TGFa-DNRII and NGFR transduced TILs and safety of treating patients with genetically modified T cells will be assessed. Feasibility will be defined as the production of virally transduced T cells and treatment of patients with these cells.
(Cohort B) The primary endpoint of growing enough TIL for patient treatment and sample size is 15 patients. | Up to 6 months
  The primary endpoint is feasibility (F) of growing enough TIL for patient treatment and sample size is 15 patients.) If you assume that Prob(F) follows 2s a non-informative beta (0.50, 0.50)prior, which has mean = 0.50 and effective sample size =1, then for example, if you observe 5/15 patients for whom F occurred and 10/15 for whom it did not, then a posterior 95% credible interval for Prob(F) would have lower and upper limits 0.14 to 0.58.

SECONDARY OUTCOMES:
(Cohort A) Response | Up to 24 months
  Will be defined following immune-related response criteria as a 50% or greater decrease in the tumor's linear dimension post treatment compared to baseline.
(Cohort A) Number of DNRII transduced cells | 6 months
  A linear regression model will be used to test the hypothesis that the DNRII cells are more likely to survive longer in the tumor environment than the NGFR (control) cells. Dose will be included as a covariate. Separate analyses will be performed at each post-treatment time point (6 weeks, 12 weeks, 6 months, 12 months, and 24 months), with the 6-month time point considered primary. If there is evidence of a linear relationship over time, a generalized linear mixed model (GLMM) approach may be used to model the DNRII/NGFR ratio over time.
(Cohort A) Number of NGFR transduced cells at infusion | Day 0
  A linear regression model will be used to test the hypothesis that the DNRII cells are more likely to survive longer in the tumor environment than the NGFR (control) cells. Dose will be included as a covariate. Separate analyses will be performed at each post-treatment time point (6 weeks, 12 weeks, 6 months, 12 months, and 24 months), with the 6-month time point considered primary. If there is evidence of a linear relationship over time, a GLMM approach may be used to model the DNRII/NGFR ratio over time.
(Cohort A) Number of NGFR transduced cells based on tumor biopsy | Up to 24 months
  A linear regression model will be used to test the hypothesis that the DNRII cells are more likely to survive longer in the tumor environment than the NGFR (control) cells. Dose will be included as a covariate. Separate analyses will be performed at each post-treatment time point (6 weeks, 12 weeks, 6 months, 12 months, and 24 months), with the 6-month time point considered primary. If there is evidence of a linear relationship over time, a GLMM approach may be used to model the DNRII/NGFR ratio over time.

CONTACTS AND LOCATIONS:
Overall Officials: Rodabe N Amaria, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org